CLINICAL TRIAL: NCT02404974
Title: Using Web-based Tools to Facilitate Tailored Exercise for People With Osteoarthritis
Acronym: exercise/OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 00028445
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Osteoarthritis
Keywords: physical activity
MeSH Terms: conditions — Osteoarthritis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise (Experimental): This is a single arm pilot study. All participants who answer yes to interest in exercise question on the web-based osteoarthritis preference tool will be included in the exercise intervention. After completing baseline measures, they will be put in contact with the Fitness Instructor and follow the protocol described.
  Interventions: Behavioral: exercise

INTERVENTIONS:
Behavioral: exercise — Participants will meet with a Certified Fitness Trainer and engage in shared goal setting and selection of a CDC-recommended exercise program for OA that best fits their needs and preferences, specifically addressing any identified barriers. The Trainer will use programs from a vetted list of programs that are appropriate for older adults with knee OA, and modify as needed. This list will be developed with the Certified Fitness Trainer and the PI. The Trainer will be available to answer questions and will contact each participant by phone every two weeks to find out how participants are doing; make adjustments to the program, if needed; and provide motivation and encouragement.

SUMMARY:
The purpose of this pilot study is to assess the feasibility, acceptability, and potential effectiveness of identifying people with osteoarthritis (OA) who are interested in individualized exercise programs through a web-based osteoarthritis application; assessing their exercise barriers, facilitators, motivators and preferences; and engaging them in an exercise program tailored to meet their needs by a Certified Fitness Trainer.

DETAILED DESCRIPTION:
The investigators hypothesize that it is feasible and acceptable to identify people with knee pain and osteoarthritis (OA) who are interested in individualized exercise programs through a web-based osteoarthritis treatment diagnosis application; to assess their exercise barriers, facilitators, motivators and preferences; and engage them in an exercise program tailored to meet their needs by a Certified Fitness Trainer.

The investigators will accomplish this by:

1. Evaluating the feasibility of identifying patients using a web-based preference diagnosis tool (PDx) who have knee pain and osteoarthritis and do not meet exercise guidelines but are interested in tailored exercise programs;
2. Evaluating the feasibility and acceptability of using self-report assessment tools to identify barriers, facilitators, motivators, and preferences for exercise and to screen participants for health problems that will limit their ability to exercise safely; and
3. Evaluating the feasibility and potential effectiveness of using the exercise assessment tool by patients with knee pain and osteoarthritis to select an individualized exercise program with the help of a Certified Fitness Trainer and to engage in routine physical exercise.

3. Study Design

Study design: The investigators will use a pre-post pilot study design. The assessments will be held at either the Dartmouth-Hitchcock Medical Center (One Medical Center Drive, Lebanon NH 03756), or The Dartmouth Centers for Health and Aging (46 Centerra Parkway, Lebanon, NH 03766). Assessments will be conducted by the principal investigator (PI), and/or a research assistant (RA). Consent and approval of the Committee for the Protections of Human Subjects of Dartmouth College will be obtained prior to starting the study. Volunteer non-exercising and under-exercising participants aged 50-85 will be recruited through flyers and provider referral. Recruitment will continue until 10 participants answer "yes" to the exercise question on PDx. Written informed consent will be obtained for all participants.

Aim 1 Methods: Feasibility of identifying patients using a web-based preference diagnosis tool (PDx) who have knee pain and osteoarthritis and do not exercise at recommended levels but are interested in tailored exercise programs.

Volunteer participants will be screened by the RA for eligibility for the study. Demographics of age and sex will be recorded at screening. After obtaining written informed consent, each eligible participant will complete the Preference Diagnosis (PDx) web-based software program and respond "yes" or "no" to the question "I am interested in an exercise program tailored to meet my needs" at the end of the program. PDx is a software application under development at The Dartmouth Center for Health Care Delivery Science (TDC) that uses weighted values and patient assessments of perceived unfavorable aspects or "costs", versus perceived benefits, to develop a profile of preferences around knee OA treatment. An RA (trained by Catalina Gorla of TDC to administer PDx) will coach participants through using the PDx program which will be administered on a lap top computer in a private room. All participants will have their height, weight, and waist circumference measured prior to starting the application using a standardized protocol. Feasibility will be assessed by the proportion of potentially eligible participants who endorse the exercise question within a 3-month period until a maximum of 10 is reached.

Aim 2 Methods: Feasibility and acceptability of using a self-report assessment to identify barriers, facilitators, motivators, and preferences for exercise and to screen participants for health problems that will limit their ability to exercise safely.

Participants who answer "yes" to the exercise question (the final question of the tool) will immediately complete a self-report screening tool: Exercise Barriers, Facilitators, Motivators, and Preferences in Older Adults (appendix A).24 The exercise assessment tool is currently under iterative development and will incorporate expertise of the Certified Fitness Trainer. Participants who are age 69 or less will also complete Personal Assessment of Readiness Questionnaire (PAR-Q) (appendix B).21 As PAR-Q is not validated in adults over 69 years, participants who answer yes to any of the questions (with the excpetion of question 5) on the PAR-Q and those older than 69 will complete a medical screening prior to participation in exercise portion of the study. If question 5 (Do you have any bone or joint problem (for example, back, knee or hip) that could be made worse by a change in your physical activity?) on the PAR-Q is endorsed, the following questions will be asked:

1. Do you have a bone or joint problem other than osteoarthritis of the knee? If no, then they will be allowed to participate in the study; If yes, they will be asked:
2. Do you have inflammatory arthritis such as Rheumatoid Arthritis, Psoriatic Arthritis, Gout, or Infectious Arthritis, such as Lyme disease? If yes, they will be excluded from participation.
3. If uncertain, they will be referred for medical screening prior to participation.

The RA will assist participants in completing assessments, if needed, and help arrange medical follow up. Feasibility will be assessed by the proportion of participants who answered "yes" to the exercise question who complete the Barriers, Facilitators, Motivators and Preferences screening and the PAR-Q and/or medical screening. Acceptability will be assessed by qualitative semi-structured one-hour interviews of the 10 participants at 3 months that will be conducted by the RA based upon questions developed by the research team (Appendix D). Interviews will be transcribed, de-indentified, coded and analyzed for themes using grounded theory.

Aim 3 Methods: Feasibility and potential effectiveness of using the self-report exercise assessment by patients with knee pain and OA to select an individualized exercise program and engage in routine physical exercise with the support of a Certified Fitness Trainer.

Participants will meet with a Certified Fitness Trainer and engage in shared goal setting and selection of a CDC-recommended exercise program for OA that best fits their needs and preferences, specifically addressing any identified barriers. The Trainer will use programs from a vetted list of programs that are appropriate for older adults with knee OA, and modify as needed. This list will be developed with the Certified Fitness Trainer and the PI. The Trainer will be available to answer questions and will contact each participant by phone every two weeks to find out how participants are doing; make adjustments to the program, if needed; and provide motivation and encouragement. Feasibility will be evaluated by quantifying the proportion of participants who complete the assessments within a 3-month period. Potential effectiveness will be evaluated based on pre-post difference in the mean number of self-reported minutes spent in mild, moderate, or vigorous exercise in the previous week; the proportion of participants who have adopted any exercise routine, and change in health goal attainment confidence. Pain as measured on a 10 cm visual analog scale will be collected as an exploratory measure. (see descriptions of measures below).

ELIGIBILITY:
Inclusion Criteria:

* Exercise <150 minutes a week of mild-moderate activity or < 75 minutes a week of vigorous activity;
* Age ≥ 50 and ≤ 85;
* Self-reported uni- or bilateral knee pain in the past 12 months that has been diagnosed as osteoarthritis and is not due to an acute injury;
* Ability to speak and read English; and
* Have an established relationship with a Primary Care Provider.

Exclusion Criteria:

* Exercise ≥150 minutes a week of mild-moderate activity or ≥ 75 minutes a week of vigorous activity;
* Age < 50 years or > 85;
* Unable to speak and read English;
* Demonstrate a profound hearing or cognitive impairment;
* Bilateral knee replacements;
* Health reasons that preclude their participation in the study such as, but not limited to, traumatic knee injury within the past 12 months, rheumatoid or other inflammatory arthritis, unstable angina, uncompensated heart failure, or their health care provider's recommendation that they not participate; or
* No established Primary Care Provider.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants completing PDx and endorsing the exercise question | 3 months
  We will record the number of participants who endorse the exercise question over the number of participants who complete PDx

SECONDARY OUTCOMES:
mean minutes of exercise | 1 and 3 months
  change in mean number of minutes spent in mild, moderate and vigorous exercise
RAPA | 1 and 3 months
  change in the Rapid Assessment of Physical Activity (RAPA) at 1 and 3 months
confidence as measured on a visual analog scale | 1 and 3 months
  Change in confidence to manage health problems as measured on a visual analog scale
Pain as measured by the 10 cm visual analog pain scale | 1 and 3 months
  change in 10 cm visual analog pain scale measured at 1 and 3 months

OTHER OUTCOMES:
qualitative analysis | 3 months
  Semistructured interviews of participants regarding acceptability of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alicia J Zbehlik, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No